CLINICAL TRIAL: NCT00993447
Title: Immunogenicity and Safety of Sanofi Pasteur's CYD Dengue Vaccine in Healthy Children and Adolescents Aged 9 to 16 Years in Latin America
Brief Title: Immunogenicity and Safety of Sanofi Pasteur's CYD Dengue Vaccine in Healthy Children and Adolescents in Latin America
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CYD13; UTN: U1111-1111-5511
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Hemorrhagic Fever; Dengue Virus; Dengue Fever
Keywords: Dengue; Dengue hemorrhagic fever; Dengue virus; Dengue fever; Sanofi pasteur's CYD Dengue vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dengue Vaccines; adacel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Sanofi pasteur's CYD Dengue vaccine group (Dengvaxia®)
  Interventions: Biological: CYD Dengue Vaccine
- Control Vaccine Group (Sham Comparator)
  Interventions: Biological: Tetanus Toxoid Reduced Diphtheria Toxoid Acellular Pertussis

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous at Day 0, 6 and 12 months
  Other Names: Dengvaxia®
  Arms: CYD Dengue Vaccine Group
Biological: Tetanus Toxoid Reduced Diphtheria Toxoid Acellular Pertussis — NaCl: 0.5 mL, Intramuscular at Day 0 and 6 months; Adacel®: 0.5 mL, Intramuscular at 12 months
  Other Names: ADACEL®; NaCl
  Arms: Control Vaccine Group

SUMMARY:
Primary objectives:

* To describe the immune response to each dengue serotype before and after each vaccination with sanofi pasteur's CYD dengue vaccine.
* To evaluate the safety of each vaccination with sanofi pasteur's CYD dengue vaccine.

DETAILED DESCRIPTION:
The antibody levels against each serotype will be measured before and after each vaccination. The subjects will be followed for 28 days after each vaccination for solicited and unsolicited safety parameters. Serious adverse events (SAEs) will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria :

* Aged 9 to 16 years on the day of inclusion
* Subject in good health, based on medical history and physical examination
* Provision of assent form/informed consent form signed by the subject and by the parent(s) or another legally acceptable representative
* Subject and parent(s)/legally acceptable representative(s) able to attend all scheduled visits and to comply with all trial procedures
* For a female subject of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to first vaccination until at least 4 weeks after the last vaccination.

Exclusion Criteria :

* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia
* For a female subject of child-bearing potential, known pregnancy or positive urine pregnancy test at Visit 1
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Breast-feeding woman
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the components of any of the trial vaccines or history of a life-threatening reaction to any of the trial vaccines or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the preceding 3 months that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination
* Subject deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* Severe diseases with or without fever, convulsions or neurological abnormalities without treatment or in progression.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Bucaramanga, Colombia
- Tegucigalpa, Honduras
- Cuernavaca, Mexico
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Villar LA, Rivera-Medina DM, Arredondo-Garcia JL, Boaz M, Starr-Spires L, Thakur M, Zambrano B, Miranda MC, Rivas E, Dayan GH. Safety and immunogenicity of a recombinant tetravalent dengue vaccine in 9-16 year olds: a randomized, controlled, phase II trial in Latin America. Pediatr Infect Dis J. 2013 Oct;32(10):1102-9. doi: 10.1097/INF.0b013e31829b8022. PMID 24067553
- [Derived] Coronel D, Garcia-Rivera EJ, Rivera DM, Arredondo-Garcia JL, Dietze R, Perroud AP, Cortes M, Bonaparte M, Wang H, Pagnon A, Jantet-Blaudez F, Penalosa LAR, Dayan G, Zambrano B, DiazGranados CA, Noriega F. Immune Response Persistence and Safety of a Booster Dose of the Tetravalent Dengue Vaccine in Adolescents and Adults Who Previously Completed the 3-dose Schedule 4-5 Years Earlier in Latin America: A Randomized Placebo-controlled Trial. Pediatr Infect Dis J. 2020 Oct;39(10):961-968. doi: 10.1097/INF.0000000000002830. PMID 32932330
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 09 October 2009 to 25 February 2010 in 3 clinic centers in Colombia, 1 in Honduras, 3 in Mexico, and 1 in Puerto Rico.
Pre-assignment Details: A total of 600 participants who met all inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Dengue Vaccine Group: Participants received the 5555 formulation of Sanofi Pasteur's CYD dengue vaccine as first (Day 0), second (Day 0 + 6 months), and third (Day 0 + 12 months) injections.
- Control Group: Participants received a placebo (NaCl) as first (Day 0) and second (Day 0 + 6 months) injections and ADACEL vaccine as a third (Day 0 + 12 months) injection.
Period: Overall Study
Arm/Group | Dengue Vaccine Group | Control Group
Started | 401 | 199
Completed | 364 | 180
Not Completed | 37 | 19
Not completed — Withdrawal by Subject | 23 | 8
Not completed — Protocol Violation | 12 | 8
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 401 | 199 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 401 | 199 | 600
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.6 (2.1) | 12.5 (2.1) | 12.55 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 108 | 312
  Male | 197 | 91 | 288
Region of Enrollment [Number; unit: Participants]
  Colombia | 105 | 54 | 159
  Honduras | 106 | 52 | 158
  Mexico | 119 | 58 | 177
  Puerto Rico | 71 | 35 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers of ≥10 1/Dil Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT).
Time Frame: Day 0 (pre-each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 401 | 199
Percentage of participants
  Serotype 1; Pre-inj. 1 (N=379,191) | 64.9 | 68.1
  Serotype 1; Post-inj. 1 (N=379,191) | 73.1 | 67.0
  Serotype 1; Pre-inj. 2 (N=353,174) | 75.6 | 67.8
  Serotype 1; Post-inj. 2 (N=353,174) | 85.0 | 69.0
  Serotype 1; Pre-inj. 3 (N=335,163) | 79.7 | 73.6
  Serotype 1; Post-inj. 3 (N=335,163) | 94.6 | 75.5
  Serotype 2; Pre-inj. 1 (N=379,191) | 69.9 | 74.3
  Serotype 2; Post-inj. 1 (N=379,191) | 85.2 | 72.8
  Serotype 2; Pre-inj. 2 (N=353,174) | 87.3 | 71.8
  Serotype 2; Post-inj. 2 (N=353,174) | 96.9 | 73.0
  Serotype 2; Pre-inj. 3 (N=335,163) | 91.9 | 76.7
  Serotype 2; Post-inj. 3 (N=335,163) | 99.1 | 78.5
  Serotype 3; Pre-inj. 1 (N=379,191) | 69.9 | 73.3
  Serotype 3; Post-inj. 1 (N=379,191) | 90.8 | 74.3
  Serotype 3; Pre-inj. 2 (N=353,174) | 90.9 | 72.4
  Serotype 3; Post-inj. 2 (N=353,174) | 98.6 | 73.6
  Serotype 3; Pre-inj. 3 (N=335,163) | 96.4 | 74.8
  Serotype 3; Post-inj. 3 (N=335,163) | 100.0 | 76.7
  Serotype 4; Pre-inj. 1 (N=379,191) | 63.1 | 68.1
  Serotype 4; Post-inj. 1 (N=379,191) | 92.6 | 62.3
  Serotype 4; Pre-inj. 2 (N=353,174) | 92.4 | 66.7
  Serotype 4; Post-inj. 2 (N=353,174) | 96.6 | 70.1
  Serotype 4; Pre-inj. 3 (N=335,163) | 95.8 | 69.9
  Serotype 4; Post-inj. 3 (N=335,163) | 98.8 | 69.3

2. Primary Outcome: Percentage of Flavi Virus-Immune Participants at Baseline With Antibody Titers ≥10 1/Dil Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Flavi virus (FV) immune participants at baseline are defined as those participants with ≥ 10 1/dil for at least one serotype with the parental dengue virus strain or for Yellow Fever titer.
Time Frame: Day 0 (pre-each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 316 | 160
Percentage of Participants
  Serotype 1; Pre-inj. 1 (N=316,160) | 81.3 | 84.4
  Serotype 1; Post-inj. 1 (N=305,158) | 90.8 | 82.3
  Serotype 1; Pre-inj. 2 (N=295,148) | 90.5 | 82.4
  Serotype 1; Post-inj. 2 (N=293,147) | 95.6 | 84.4
  Serotype 1; Pre-inj. 3 (N=288,143) | 92.0 | 87.4
  Serotype 1; Post-inj. 3 (N=287,143) | 97.6 | 88.8
  Serotype 2; Pre-inj. 1 (N=316,160) | 88.0 | 91.9
  Serotype 2; Post-inj. 1 (N=305,158) | 96.4 | 89.9
  Serotype 2; Pre-inj. 2 (N=295,148) | 96.6 | 89.2
  Serotype 2; Post-inj. 2 (N=293,147) | 98.6 | 90.5
  Serotype 2; Pre-inj. 3 (N=288,143) | 96.5 | 90.9
  Serotype 2; Post-inj. 3 (N=287,143) | 99.7 | 92.3
  Serotype 3; Pre-inj. 1 (N=316,160) | 88.3 | 90.6
  Serotype 3; Post-inj. 1 (N=305,158) | 96.7 | 89.9
  Serotype 3; Pre-inj. 2 (N=295,148) | 96.6 | 87.8
  Serotype 3; Post-inj. 2 (N=293,147) | 99.0 | 88.4
  Serotype 3; Pre-inj. 3 (N=288,143) | 97.9 | 89.5
  Serotype 3; Post-inj. 3 (N=287,143) | 100.0 | 89.5
  Serotype 4; Pre-inj. 1 (N=316,160) | 79.4 | 84.4
  Serotype 4; Post-inj. 1 (N=305,158) | 97.4 | 76.6
  Serotype 4; Pre-inj. 2 (N=295,148) | 96.9 | 81.1
  Serotype 4; Post-inj. 2 (N=293,147) | 98.0 | 84.4
  Serotype 4; Pre-inj. 3 (N=288,143) | 99.3 | 84.6
  Serotype 4; Post-inj. 3 (N=287,143) | 100.0 | 84.6

3. Primary Outcome: Percentage of Flavi Virus-Naive Participants at Baseline With Antibody Titers ≥10 1/Dil Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Flavi virus (FV) naïve participants are defined as those participants with < 10 1/dil for all serotypes with parental dengue virus strains and for Yellow Fever titer.
Time Frame: Day 0 (pre-each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 85 | 38
Percentage of participants
  Serotype 1; Pre-inj. 1 (N=85,38) | 0.0 | 0.0
  Serotype 1; Post-inj. 1 (N=84,37) | 7.1 | 2.7
  Serotype 1; Pre-inj. 2 (N=78,36) | 17.9 | 5.6
  Serotype 1; Post-inj. 2 (N=78,36) | 44.9 | 5.6
  Serotype 1; Pre-inj. 3 (N=77,36) | 33.8 | 16.7
  Serotype 1; Post-inj. 3 (N=77,36) | 81.8 | 19.4
  Serotype 2; Pre-inj. 1 (N=85,38) | 0.0 | 0.0
  Serotype 2; Post-inj. 1 (N=84,37) | 42.9 | 0.0
  Serotype 2; Pre-inj. 2 (N=78,36) | 51.3 | 2.8
  Serotype 2; Post-inj. 2 (N=78,36) | 89.7 | 5.6
  Serotype 2; Pre-inj. 3 (N=77,36) | 70.1 | 16.7
  Serotype 2; Post-inj. 3 (N=77,36) | 96.1 | 19.4
  Serotype 3; Pre-inj. 1 (N=85,38) | 0.0 | 0.0
  Serotype 3; Post-inj. 1 (N=84,37) | 67.9 | 10.8
  Serotype 3; Pre-inj. 2 (N=78,36) | 66.7 | 8.3
  Serotype 3; Post-inj. 2 (N=78,36) | 94.9 | 8.3
  Serotype 3; Pre-inj. 3 (N=77,36) | 89.6 | 5.6
  Serotype 3; Post-inj. 3 (N=77,36) | 100.0 | 16.7
  Serotype 4; Pre-inj. 1 (N=85,38) | 0.0 | 0.0
  Serotype 4; Post-inj. 1 (N=84,37) | 73.8 | 2.7
  Serotype 4; Pre-inj. 2 (N=78,36) | 73.1 | 5.6
  Serotype 4; Post-inj. 2 (N=78,36) | 91.0 | 8.3
  Serotype 4; Pre-inj. 3 (N=77,36) | 80.5 | 8.3
  Serotype 4; Post-inj. 3 (N=77,36) | 94.8 | 5.6

4. Primary Outcome: Percentage of Participants With Antibody Titers of ≥10 1/Dil Against At Least 1, 2, 3, or 4 Serotypes With Parental Dengue Virus Strain Before and Following Each Injection With Either Sanofi Pasteur's CYD Dengue Vaccine or A Placebo Vaccine
Description: as for outcome 1
Time Frame: Day 0 (before each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Per Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 401 | 199
Percentage of participants
  At Least 1 Serotype; Pre-inj 1; 1 (N=401,199) | 75.1 | 77.9
  At Least 1 Serotype; Post-inj. 1 (N=389,196) | 98.2 | 78.6
  At Least 1 Serotype; Pre-inj. 2 (N=373,185) | 99.2 | 76.2
  At Least 1 Serotype; Post-inj. 2 (N=371,184) | 99.7 | 76.6
  At Least 1 Serotype; Pre-inj. 3 (N=365,180) | 100.0 | 79.4
  At Least 1 Serotype; Post-inj. 3 (N=364,180) | 100.0 | 78.9
  At Least 2 Serotypes; Pre-inj. 1 (N=401,199) | 69.1 | 72.9
  At Least 2 Serotypes; Post-inj. 1 (N=389,196) | 91.0 | 70.9
  At Least 2 Serotypes; Pre-inj. 2 (N=373,185) | 91.4 | 71.9
  At Least 2 Serotypes; Post-inj. 2 (N=371,184) | 98.9 | 71.2
  At Least 2 Serotypes; Pre-inj. 3 (N=365,180) | 96.2 | 75.6
  At Least 2 Serotypes; Post-inj. 3 (N=364,180) | 100.0 | 76.7
  At Least 3 Serotypes; Pre-inj. 1 (N=401,199) | 64.6 | 69.8
  At Least 3 Serotypes; Post-inj. 1 (N=381,196) | 79.9 | 67.3
  At Least 3 Serotypes; Pre-inj. 2 (N=373,185) | 81.8 | 68.1
  At Least 3 Serotypes; Post-inj. 2 (N=371,184) | 94.3 | 69.0
  At Least 3 Serotypes; Pre-inj. 3 (N=365,180) | 88.2 | 70.6
  At Least 3 Serotypes; Post-inj. 3 (N=364,180) | 98.6 | 72.2
  All 4 Serotypes; Pre-inj. 1 (N=401,199) | 56.9 | 61.8
  All 4 Serotypes; Post-inj. 1 (N=389,196) | 71.2 | 59.2
  All 4 Serotypes; Pre-inj. 2 (N=373,185) | 72.4 | 60.5
  All 4 Serotypes; Post-inj. 2 (N=371,184) | 83.3 | 66.3
  All 4 Serotypes; Pre-inj. 3 (N=365,180) | 77.8 | 64.4
  All 4 Serotypes; Post-inj. 3 (N=364,180) | 93.4 | 66.7

5. Primary Outcome: Percentage of Flavi Virus-Immune Participants With Antibody Titers of ≥10 1/Dil Against At Least 1, 2, 3, or 4 Serotypes With Parental Dengue Virus Strain Pre and Post-Injection With Either Sanofi Pasteur's CYD Dengue Vaccine or A Placebo Vaccine
Description: as for outcome 1
Time Frame: Day 0 (before each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Per Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 316 | 160
Percentage of participants
  At Least 1 Serotype; Pre-inj 1; 1 (N=401,199) | 95.3 | 96.9
  At Least 1 Serotype; Post-inj. 1 (N=389,196) | 99.0 | 93.7
  At Least 1 Serotype; Pre-inj. 2 (N=373,185) | 99.7 | 91.9
  At Least 1 Serotype; Post-inj. 2 (N=371,184) | 99.7 | 93.2
  At Least 1 Serotype; Pre-inj. 3 (N=365,180) | 100.0 | 93.7
  At Least 1 Serotype; Post-inj. 3 (N=364,180) | 100.0 | 93.0
  At Least 2 Serotypes; Pre-inj. 1 (N=401,199) | 87.7 | 90.6
  At Least 2 Serotypes; Post-inj. 1 (N=389,196) | 97.4 | 88.0
  At Least 2 Serotypes; Pre-inj. 2 (N=373,185) | 97.3 | 89.2
  At Least 2 Serotypes; Post-inj. 2 (N=371,184) | 99.0 | 87.8
  At Least 2 Serotypes; Pre-inj. 3 (N=365,180) | 98.6 | 91.6
  At Least 2 Serotypes; Post-inj. 3 (N=364,180) | 100.0 | 92.3
  At Least 3 Serotypes; Pre-inj. 1 (N=401,199) | 92.0 | 86.9
  At Least 3 Serotypes; Post-inj. 1 (N=381,196) | 95.1 | 83.5
  At Least 3 Serotypes; Pre-inj. 2 (N=373,185) | 94.2 | 84.5
  At Least 3 Serotypes; Post-inj. 2 (N=371,184) | 98.3 | 85.0
  At Least 3 Serotypes; Pre-inj. 3 (N=365,180) | 96.2 | 86.7
  At Least 3 Serotypes; Post-inj. 3 (N=364,180) | 99.7 | 87.4
  All 4 Serotypes; Pre-inj. 1 (N=401,199) | 72.2 | 76.9
  All 4 Serotypes; Post-inj. 1 (N=389,196) | 89.8 | 73.4
  All 4 Serotypes; Pre-inj. 2 (N=373,185) | 89.5 | 75.0
  All 4 Serotypes; Post-inj. 2 (N=371,184) | 94.2 | 81.6
  All 4 Serotypes; Pre-inj. 3 (N=365,180) | 91.0 | 80.4
  All 4 Serotypes; Post-inj. 3 (N=364,180) | 97.6 | 82.5

6. Primary Outcome: Percentage of Flavi Virus-Naive Participants With Antibody Titers of ≥10 1/Dil Against At Least 1, 2, 3, or 4 Serotypes With Parental Dengue Virus Strain Pre and Post-Injection With Either Sanofi Pasteur's CYD Dengue Vaccine or A Placebo Vaccine
Description: as for outcome 1
Time Frame: Day 0 (before each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Per Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 85 | 38
Percentage of participants
  At Least 1 Serotype; Pre-inj 1; 1 (N=401,199) | 0.0 | 0.0
  At Least 1 Serotype; Post-inj. 1 (N=389,196) | 95.0 | 16.2
  At Least 1 Serotype; Pre-inj. 2 (N=373,185) | 97.4 | 13.9
  At Least 1 Serotype; Post-inj. 2 (N=371,184) | 100.0 | 11.1
  At Least 1 Serotype; Pre-inj. 3 (N=365,180) | 100.0 | 22.2
  At Least 1 Serotype; Post-inj. 3 (N=364,180) | 100.0 | 25.0
  At Least 2 Serotypes; Pre-inj. 1 (N=401,199) | 0.0 | 0.0
  At Least 2 Serotypes; Post-inj. 1 (N=389,196) | 67.9 | 0.0
  At Least 2 Serotypes; Pre-inj. 2 (N=373,185) | 69.2 | 2.8
  At Least 2 Serotypes; Post-inj. 2 (N=371,184) | 98.7 | 5.6
  At Least 2 Serotypes; Pre-inj. 3 (N=365,180) | 87.0 | 13.9
  At Least 2 Serotypes; Post-inj. 3 (N=364,180) | 100.0 | 16.7
  At Least 3 Serotypes; Pre-inj. 1 (N=401,199) | 0.0 | 0.0
  At Least 3 Serotypes; Post-inj. 1 (N=381,196) | 25.0 | 0.0
  At Least 3 Serotypes; Pre-inj. 2 (N=373,185) | 34.6 | 2.8
  At Least 3 Serotypes; Post-inj. 2 (N=371,184) | 79.5 | 5.6
  At Least 3 Serotypes; Pre-inj. 3 (N=365,180) | 58.4 | 8.3
  At Least 3 Serotypes; Post-inj. 3 (N=364,180) | 94.8 | 13.9
  All 4 Serotypes; Pre-inj. 1 (N=401,199) | 0.0 | 0.0
  All 4 Serotypes; Post-inj. 1 (N=389,196) | 3.6 | 0.0
  All 4 Serotypes; Pre-inj. 2 (N=373,185) | 7.7 | 2.8
  All 4 Serotypes; Post-inj. 2 (N=371,184) | 42.3 | 5.6
  All 4 Serotypes; Pre-inj. 3 (N=365,180) | 28.6 | 2.8
  All 4 Serotypes; Post-inj. 3 (N=364,180) | 77.9 | 5.6

7. Primary Outcome: Summary of Geometric Mean Titers (GMTs) of Antibodies Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: as for outcome 1
Time Frame: Day 0 (before each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 401 | 199
Titers (1/dilution)
  Serotype 1; Pre-inj. 1 (N=401,199) | 74.2 [58.8 to 93.6] | 81.9 [59.2 to 113]
  Serotype 1; Post-inj. 1 (N=389,196) | 221 [167 to 292] | 77.1 [55.8 to 106]
  Serotype 1; Pre-inj. 2 (N=373,185) | 193 [149 to 251] | 96.6 [67.1 to 139]
  Serotype 1; Post-inj. 2 (N=371,184) | 276 [215 to 355] | 102 [70.9 to 147]
  Serotype 1; Pre-inj. 3 (N=365,180) | 204 [159 to 262] | 113 [80.0 to 159]
  Serotype 1; Post-inj. 3 (N=364,180) | 320 [258 to 396] | 106 [75.4 to 149]
  Serotype 2; Pre-inj. 1 (N=401,199) | 92.6 [73.9 to 116] | 100 [73.5 to 136]
  Serotype 2; Post-inj. 1 (N=389,196) | 409 [320 to 524] | 90.4 [66.6 to 123]
  Serotype 2; Pre-inj. 2 (N=373,185) | 326 [260 to 408] | 117 [82.2 to 166]
  Serotype 2; Post-inj. 2 (N=371,184) | 504 [414 to 613] | 114 [80.8 to 160]
  Serotype 2; Pre-inj. 3 (N=365,180) | 300 [245 to 368] | 133 [95.6 to 186]
  Serotype 2; Post-inj. 3 (N=364,180) | 486 [414 to 572] | 133 [96.2 to 185]
  Serotype 3; Pre-inj. 1 (N=401,199) | 85.0 [68.1 to 106] | 88.8 [65.9 to 120]
  Serotype 3; Post-inj. 1 (N=389,196) | 442 [352 to 554] | 93.2 [69.1 to 126]
  Serotype 3; Pre-inj. 2 (N=372,185) | 301 [243 to 372] | 107 [77.0 to 149]
  Serotype 3; Post-inj. 2 (N=371,184) | 502 [421 to 599] | 108 [76.8 to 151]
  Serotype 3; Pre-inj. 3 (N=365,180) | 379 [313 to 458] | 123 [87.3 to 172]
  Serotype 3; Post-inj. 3 (N=364,180) | 594 [511 to 692] | 121 [86.6 to 168]
  Serotype 4; Pre-inj. 1 (N=401,199) | 37.2 [31.1 to 44.5] | 40.1 [31.2 to 51.5]
  Serotype 4; Post-inj. 1 (N=389,196) | 416 [347 to 498] | 34.1 [26.5 to 43.9]
  Serotype 4; Pre-inj. 2 (N=373,185) | 200 [171 to 233] | 43.8 [33.2 to 57.8]
  Serotype 4; Post-inj. 2 (N=369,184) | 305 [265 to 352] | 43.9 [33.5 to 57.5]
  Serotype 4; Pre-inj. 3 (N=365,180) | 182 [158 to 210] | 47.7 [36.4 to 62.6]
  Serotype 4; Post-inj. 3 (N=364,180) | 273 [241 to 309] | 42.8 [33.0 to 55.5]

8. Primary Outcome: Summary of Geometric Mean Titers Ratios of Antibodies Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Geometric mean titer ratio is the geometric mean of individual post vaccination/pre vaccination titer of antibodies to each parental dengue virus serotype strain.
Time Frame: Day 0 (before each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 401 | 199
Titers
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=389,196) | 2.36 [2.02 to 2.76] | 0.756 [0.689 to 0.829]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=371,184) | 2.74 [2.33 to 3.21] | 1.02 [0.820 to 1.27]
  Serotype 1; Post-inj. 2/Pre-inj. 2 (N=371,184) | 1.19 [1.06 to 1.34] | 0.851 [0.735 to 0.985]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=364,180) | 3.16 [2.73 to 3.66] | 1.03 [0.834 to 1.27]
  Serotype 1; Post-inj. 3/Pre-inj. 2 (N=364,180) | 1.38 [1.22 to 1.56] | 0.859 [0.710 to 1.04]
  Serotype 1; Post-inj. 3/Pre-inj. 3 (N=364,180) | 1.35 [1.25 to 1.46] | 0.777 [0.699 to 0.862]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=389,196) | 3.55 [3.04 to 4.15] | 0.760 [0.702 to 0.823]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=371,184) | 4.09 [3.49 to 4.80] | 0.983 [0.805 to 1.20]
  Serotype 2; Post-inj. 2/Pre-inj. 2 (N=371,184) | 1.40 [1.25 to 1.58] | 0.811 [0.698 to 0.941]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=364,180) | 3.97 [3.39 to 4.64] | 1.16 [0.955 to 1.41]
  Serotype 2; Post-inj. 3/Pre-inj. 2 (N=364,180) | 1.36 [1.19 to 1.55] | 0.957 [0.777 to 1.18]
  Serotype 2; Post-inj. 3/Pre-inj. 3 (N=364,180) | 1.51 [1.38 to 1.64] | 0.844 [0.770 to 0.926]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=389,196) | 4.24 [3.61 to 4.98] | 0.864 [0.786 to 0.950]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=371,184) | 4.52 [3.88 to 5.26] | 1.04 [0.852 to 1.28]
  Serotype 3; Post-inj. 2/Pre-inj. 2 (N=370,184) | 1.57 [1.40 to 1.76] | 0.840 [0.725 to 0.975]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=364,180) | 5.27 [4.55 to 6.10] | 1.15 [0.960 to 1.39]
  Serotype 3; Post-inj. 3/Pre-inj. 2 (N=363,180) | 1.86 [1.64 to 2.10] | 0.937 [0.780 to 1.13]
  Serotype 3; Post-inj. 3/Pre-inj. 3 (N=364,180) | 1.52 [1.41 to 1.63] | 0.815 [0.743 to 0.895]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=389,196) | 8.63 [7.09 to 10.5] | 0.672 [0.603 to 0.750]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=369,184) | 6.14 [5.22 to 7.21] | 0.887 [0.725 to 1.09]
  Serotype 4; Post-inj. 2/Pre-inj. 2 (N=369,184) | 1.45 [1.29 to 1.62] | 0.800 [0.703 to 0.911]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=364,180) | 5.47 [4.72 to 6.34] | 0.871 [0.720 to 1.05]
  Serotype 4; Post-inj. 3/Pre-inj. 2 (N=364,180) | 1.30 [1.16 to 1.46] | 0.771 [0.656 to 0.906]
  Serotype 4; Post-inj. 3/Pre-inj. 3 (N=364,180) | 1.45 [1.34 to 1.56] | 0.723 [0.671 to 0.780]

9. Primary Outcome: Summary of Geometric Mean Titers (GMTs) of Antibodies in Flavivirus-Immune Participants at Baseline Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Flavivirus-immune subjects at baseline are defined as those participants with ≥ 10 1/dil for at least one serotype with the parental dengue virus strain or for Yellow Fever titer.
Time Frame: Day 0 (before each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 316 | 160
Titers (1/dilution)
  Serotype 1; Pre-inj. 1 (N=316,160) | 153 [121 to 194] | 162 [117 to 224]
  Serotype 1; Post-inj. 1 (N=305,158) | 604 [468 to 780] | 148 [107 to 205]
  Serotype 1; Pre-inj. 2 (N=295,148) | 447 [352 to 567] | 192 [133 to 279]
  Serotype 1; Post-inj. 2 (N=293,147) | 607 [483 to 764] | 199 [138 to 287]
  Serotype 1; Pre-inj. 3 (N=288,143) | 435 [344 to 550] | 225 [161 to 315]
  Serotype 1; Post-inj. 3 (N=287,143) | 580 [471 to 715] | 205 [146 to 287]
  Serotype 2; Pre-inj. 1 (N=316,160) | 203 [164 to 252] | 207 [156 to 275]
  Serotype 2; Post-inj. 1 (N=305,158) | 1001 [811 to 1236] | 181 [136 to 242]
  Serotype 2; Pre-inj. 2 (N=295,148) | 673 [555 to 817] | 251 [179 to 351]
  Serotype 2; Post-inj. 2 (N=293,147) | 888 [738 to 1067] | 232 [167 to 321]
  Serotype 2; Pre-inj. 3 (N=288,143) | 554 [461 to 667] | 265 [195 to 361]
  Serotype 2; Post-inj. 3 (N=287,143) | 741 [631 to 869] | 266 [196 to 359]
  Serotype 3; Pre-inj. 1 (N=316,160) | 182 [147 to 225] | 179 [136 to 237]
  Serotype 3; Post-inj. 1 (N=305,158) | 863 [700 to 1064] | 180 [135 to 239]
  Serotype 3; Pre-inj. 2 (N=295,148) | 556 [456 to 679] | 221 [161 to 304]
  Serotype 3; Post-inj. 2 (N=293,147) | 782 [654 to 936] | 215 [155 to 297]
  Serotype 3; Pre-inj. 3 (N=288,143) | 615 [510 to 743] | 265 [193 to 362]
  Serotype 3; Post-inj. 3 (N=287,143) | 827 [704 to 972] | 248 [181 to 340]
  Serotype 4; Pre-inj. 1 (N=316,160) | 63.8 [52.9 to 76.9] | 66.5 [51.4 to 86.1]
  Serotype 4; Post-inj. 1 (N=305,158) | 549 [465 to 649] | 53.4 [40.8 to 69.8]
  Serotype 4; Pre-inj. 2 (N=295,148) | 278 [239 to 322] | 73.7 [55.2 to 98.5]
  Serotype 4; Post-inj. 2 (N=291,147) | 395 [341 to 456] | 70.4 [53.3 to 92.8]
  Serotype 4; Pre-inj. 3 (N=288,143) | 259 [227 to 296] | 81.8 [62.1 to 108]
  Serotype 4; Post-inj. 3 (N=287,143) | 341 [299 to 388] | 72.5 [55.8 to 94.2]

10. Primary Outcome: Summary of Geometric Mean Titers Ratios of Antibodies in Flavivirus-Immune Participants at Baseline Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Flavivirus-immune subjects at baseline are defined as those participants with ≥ 10 1/dil for at least one serotype with the parental dengue virus strain or for Yellow Fever titer. Geometric mean titer ratio is the geometric mean of individual post vaccination/pre-vaccination titer of antibodies to each parental dengue virus serotype strain.
Time Frame: Day 0 (pre each vaccination) and Day 28 post each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 316 | 160
Titers
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=305,158) | 3.49 [2.94 to 4.15] | 0.829 [0.743 to 0.924]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=293,147) | 3.25 [2.73 to 3.88] | 1.11 [0.875 to 1.41]
  Serotype 1; Post-inj. 2/Pre-inj. 2 (N=293,147) | 1.25 [1.10 to 1.43] | 0.925 [0.793 to 1.08]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=287,143) | 3.08 [2.61 to 3.64] | 1.09 [0.857 to 1.39]
  Serotype 1; Post-inj. 3/Pre-inj. 2 (N=287,143) | 1.19 [1.05 to 1.35] | 0.907 [0.723 to 1.14]
  Serotype 1; Post-inj. 3/Pre-inj. 3 (N=287,143) | 1.24 [1.15 to 1.34] | 0.834 [0.736 to 0.946]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=305,158) | 4.43 [3.74 to 5.24] | 0.840 [0.766 to 0.921]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=293,147) | 3.70 [3.08 to 4.44] | 1.08 [0.863 to 1.35]
  Serotype 2; Post-inj. 2/Pre-inj. 2 (N=293,147) | 1.27 [1.12 to 1.44] | 0.865 [0.735 to 1.02]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=287,143) | 3.08 [2.59 to 3.67] | 1.23 [0.993 to 1.53]
  Serotype 2; Post-inj. 3/Pre-inj. 2 (N=287,143) | 1.06 [0.939 to 1.20] | 0.982 [0.775 to 1.25]
  Serotype 2; Post-inj. 3/Pre-inj. 3 (N=287,143) | 1.29 [1.18 to 1.40] | 0.940 [0.846 to 1.04]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=305,158) | 4.35 [3.67 to 5.15] | 0.941 [0.850 to 1.04]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=293,147) | 3.71 [3.13 to 4.39] | 1.16 [0.921 to 1.45]
  Serotype 3; Post-inj. 2/Pre-inj. 2 (N=293,147) | 1.36 [1.20 to 1.55] | 0.906 [0.779 to 1.05]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=287,143) | 3.82 [3.27 to 4.47] | 1.29 [1.05 to 1.60]
  Serotype 3; Post-inj. 3/Pre-inj. 2 (N=287,143) | 1.43 [1.27 to 1.62] | 1.03 [0.824 to 1.28]
  Serotype 3; Post-inj. 3/Pre-inj. 3 (N=287,143) | 1.31 [1.22 to 1.40] | 0.872 [0.789 to 0.963]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=305,158) | 7.40 [6.03 to 9.08] | 0.712 [0.625 to 0.812]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=291,147) | 5.16 [4.31 to 6.19] | 0.952 [0.752 to 1.20]
  Serotype 4; Post-inj. 2/Pre-inj. 2 (N=291,147) | 1.39 [1.22 to 1.57] | 0.847 [0.739 to 0.971]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=287,143) | 4.45 [3.76 to 5.26] | 0.976 [0.773 to 1.23]
  Serotype 4; Post-inj. 3/Pre-inj. 2 (N=287,143) | 1.20 [1.06 to 1.36] | 0.849 [0.698 to 1.03]
  Serotype 4; Post-inj. 3/Pre-inj. 3 (N=287,143) | 1.30 [1.21 to 1.40] | 0.796 [0.730 to 0.868]

11. Primary Outcome: Summary of Geometric Mean Titers (GMTs) of Antibodies in Flavivirus-Naïve Participants at Baseline Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT). Flavivirus-naïve participants are defined as those participants with < 10 1/dilutions for all serotypes with parental dengue virus strains and for Yellow Fever titer.
Time Frame: Day 0 (pre-each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 85 | 38
Titers (1/dilution)
  Serotype 1; Pre-inj. 1 (N=85,38) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-inj. 1 (N=84,37) | 5.72 [5.10 to 6.42] | 5.15 [4.85 to 5.47]
  Serotype 1; Pre-inj. 2 (N=78,36) | 8.16 [5.98 to 11.1] | 6.18 [4.20 to 9.11]
  Serotype 1; Post-inj. 2 (N=78,36) | 14.3 [10.0 to 20.3] | 7.29 [4.27 to 12.5]
  Serotype 1; Pre-inj. 3 (N=77,36) | 12.0 [8.48 to 16.9] | 7.93 [5.05 to 12.5]
  Serotype 1; Post-inj. 3 (N=77,36) | 34.6 [25.0 to 48.1] | 8.36 [5.31 to 13.2]
  Serotype 2; Pre-inj. 1 (N=85,38) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-inj. 1 (N=84,37) | 15.9 [11.4 to 22.3] | 5.00 [5.00 to 5.00]
  Serotype 2; Pre-inj. 2 (N=78,36) | 21.0 [14.2 to 31.1] | 5.50 [4.54 to 6.66]
  Serotype 2; Post-inj. 2 (N=78,36) | 60.0 [43.3 to 83.0] | 6.79 [4.37 to 10.6]
  Serotype 2; Pre-inj. 3 (N=77,36) | 30.3 [21.4 to 42.7] | 9.48 [5.60 to 16.1]
  Serotype 2; Post-inj. 3 (N=77,36) | 101 [77.2 to 133] | 9.45 [5.78 to 15.4]
  Serotype 3; Pre-inj. 1 (N=85,38) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-inj. 1 (N=84,37) | 38.8 [25.6 to 59.1] | 6.10 [4.89 to 7.60]
  Serotype 3; Pre-inj. 2 (N=77,36) | 28.6 [20.0 to 41.1] | 5.97 [4.75 to 7.50]
  Serotype 3; Post-inj. 2 (N=78,36) | 94.9 [70.7 to 127] | 7.07 [4.41 to 11.3]
  Serotype 3; Pre-inj. 3 (N=77,36) | 61.9 [44.4 to 86.1] | 6.18 [4.58 to 8.34]
  Serotype 3; Post-inj. 3 (N=77,36) | 174 [136 to 221] | 7.53 [5.32 to 10.7]
  Serotype 4; Pre-inj. 1 (N=85,38) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-inj. 1 (N=84,37) | 151 [89.3 to 255] | 5.30 [4.71 to 5.96]
  Serotype 4; Pre-inj. 2 (N=78,36) | 57.5 [38.8 to 85.1] | 5.48 [4.80 to 6.26]
  Serotype 4; Post-inj. 2 (N=78,36) | 117 [84.8 to 161] | 6.77 [4.64 to 9.88]
  Serotype 4; Pre-inj. 3 (N=77,36) | 48.3 [35.5 to 65.6] | 5.97 [4.87 to 7.32]
  Serotype 4; Post-inj. 3 (N=77,36) | 119 [92.0 to 153] | 5.63 [4.76 to 6.65]

12. Primary Outcome: Summary of Geometric Mean Titer Ratios of Antibodies in Flavivirus-Naive Participants at Baseline Against Each Parental Dengue Virus Serotype Strain Before and Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Neutralizing antibody levels against each of the 4 parental dengue virus strains of Sanofi Pasteur's CYD dengue vaccine constructs were measured using the dengue plaque reduction neutralization test (PRNT).
  Flavivirus-naïve participants are defined as those participants with < 10 1/dil for all serotypes with parental dengue virus strains and for Yellow Fever titer. Geometric mean titer ratio is the geometric mean of individual post-vaccination/pre-vaccination titer of antibodies to each parental dengue virus serotype strain.
Time Frame: Day 0 (pre-each vaccination) and Day 28 post-each vaccination
Population: Antibody titers against each dengue virus serotype strain were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 85 | 38
Titers
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=84,37) | 0.572 [0.510 to 0.642] | 0.515 [0.485 to 0.547]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=78,36) | 1.43 [1.00 to 2.03] | 0.729 [0.427 to 1.25]
  Serotype 1; Post-inj. 2/Pre-inj. 2 (N=78,36) | 0.990 [0.773 to 1.27] | 0.613 [0.410 to 0.917]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=77,36) | 3.46 [2.50 to 4.81] | 0.836 [0.531 to 1.32]
  Serotype 1; Post-inj. 3/Pre-inj. 2 (N=77,36) | 2.39 [1.78 to 3.22] | 0.703 [0.512 to 0.964]
  Serotype 1; Post-inj. 3/Pre-inj. 3 (N=77,36) | 1.83 [1.48 to 2.26] | 0.592 [0.519 to 0.675]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=84,37) | 1.59 [1.14 to 2.23] | 0.500 [0.500 to 0.500]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=78,36) | 6.00 [4.33 to 8.30] | 0.679 [0.437 to 1.06]
  Serotype 2; Post-inj. 2/Pre-inj. 2 (N=78,36) | 2.04 [1.50 to 2.77] | 0.630 [0.431 to 0.921]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=77,36) | 10.1 [7.72 to 13.3] | 0.945 [0.578 to 1.54]
  Serotype 2; Post-inj. 3/Pre-inj. 2 (N=77,36) | 3.40 [2.35 to 4.91] | 0.876 [0.550 to 1.40]
  Serotype 2; Post-inj. 3/Pre-inj. 3 (N=77,36) | 2.73 [2.23 to 3.33] | 0.559 [0.493 to 0.635]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=84,37) | 3.88 [2.56 to 5.91] | 0.610 [0.489 to 0.760]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=78,36) | 9.49 [7.07 to 12.7] | 0.707 [0.441 to 1.13]
  Serotype 3; Post-inj. 2/Pre-inj. 2 (N=77,36) | 2.67 [2.13 to 3.35] | 0.627 [0.402 to 0.977]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=77,36) | 17.4 [13.6 to 22.1] | 0.753 [0.532 to 1.07]
  Serotype 3; Post-inj. 3/Pre-inj. 2 (N=76,36) | 4.90 [3.68 to 6.53] | 0.668 [0.498 to 0.896]
  Serotype 3; Post-inj. 3/Pre-inj. 3 (N=77,36) | 2.61 [2.16 to 3.16] | 0.633 [0.499 to 0.805]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=84,37) | 15.1 [8.93 to 25.5] | 0.530 [0.471 to 0.596]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=78,36) | 11.7 [8.48 to 16.1] | 0.677 [0.464 to 0.988]
  Serotype 4; Post-inj. 2/Pre-inj. 2 (N=78,36) | 1.69 [1.31 to 2.17] | 0.642 [0.445 to 0.925]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=77,36) | 11.9 [9.20 to 15.3] | 0.563 [0.476 to 0.665]
  Serotype 4; Post-inj. 3/Pre-inj. 2 (N=77,36) | 1.75 [1.31 to 2.34] | 0.533 [0.441 to 0.645]
  Serotype 4; Post-inj. 3/Pre-inj. 3 (N=77,36) | 2.15 [1.74 to 2.64] | 0.499 [0.460 to 0.541]

13. Primary Outcome: Number of Participants Reporting a Solicited Injection-site or Systemic Reactions Following Each Injection With Sanofi Pasteur's CYD Dengue Vaccine
Description: Solicited Injection-site reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Fever, (Temperature) Headache, Malaise, Myalgia, and Asthenia. Grade 3 Solicited Injection-Site Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, ≥ 5 cm. Grade 3 Solicited Systemic Reactions: Fever, ≥ 39˚C; Headache, Malaise, Myalgia, and Asthenia, Significant; prevents daily activity.
Time Frame: Day 0 up to Day 14 post-each vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set, which includes all persons who received at least one dose of study vaccine.
Measure: Number; unit: Participants
Arm/Group | Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 401 | 199
Participants
  Injection-site Pain (Any dose; N=392,198) | 192 | 132
  Grade 3 Pain (Any dose; N=392,198) | 13 | 7
  Injection-site Erythema (Any dose; N=392,198) | 26 | 18
  Grade 3 Erythema (Any dose; N=392,198) | 0 | 1
  Injection-site Swelling (Any dose; N=392,198) | 20 | 16
  Grade 3 Swelling (Any dose; N=392,198) | 1 | 1
  Injection-site Pain (Post-dose 1; N=392,196) | 121 | 54
  Grade 3 Pain (Post-dose 1; N=392,196) | 6 | 2
  Injection-site Erythema (Post-dose 1; N=390,196) | 11 | 6
  Grade 3 Erythema (Post-dose 1; N=390,196) | 0 | 0
  Injection-site Swelling (Post-dose 1; N=391,196) | 8 | 5
  Grade 3 Swelling (Post-dose 1; N=391,196) | 1 | 0
  Injection-site Pain (Post-dose 2; N=373,185) | 101 | 31
  Grade Pain (Post-dose 2; N=373,185) | 7 | 0
  Injection-site Erythema (Post-dose 2; N=373,185) | 12 | 5
  Grade 3 Erythema (Post-dose 2; N=373,185) | 0 | 0
  Injection-site Swelling (Post-dose 2; N=373,185) | 8 | 2
  Grade 3 Swelling (Post-dose 2; N=373,185) | 1 | 0
  Injection-site Pain (Post-dose 3; N=364,180) | 88 | 118
  Grade 3 Pain (Post-dose 3; N=364,180) | 2 | 5
  Injection-site Erythema (Post-dose 3; N=364,180) | 8 | 16
  Grade 3 Erythema (Post-dose 3; N=364,180) | 0 | 1
  Injection-site Swelling (Post-dose 3; N=364,180) | 6 | 14
  Grade 3 Swelling (Post-dose 3; N=364,180) | 0 | 1
  Fever (Any dose; N=392;197) | 84 | 36
  Grade 3 Fever (Any dose; N=392;197) | 13 | 3
  Headache (Any dose; N=391;198) | 237 | 116
  Grade 3 Headache (Any dose; N=391;198) | 40 | 11
  Malaise (Any dose; N=390;198) | 157 | 82
  Grade 3 Malaise (Any dose; N=390;198) | 21 | 8
  Myalgia (Any dose; N=390;198) | 171 | 90
  Grade 3 Myalgia (Any dose; N=390;198) | 22 | 10
  Asthenia (Any dose; N=390;198) | 119 | 51
  Grade 3 Asthenia (Any dose; N=390;198) | 14 | 5
  Fever (Post-dose 1; N=392;193) | 43 | 13
  Grade 3 Fever (Post dose 1; N=392;193) | 11 | 0
  Headache (Post-dose 1; N=391;197) | 173 | 80
  Grade 3 Headache (Post-dose 1; N=391;197) | 26 | 5
  Malaise (Post-dose 1; N=390;197) | 102 | 45
  Grade 3 Malaise (Post-dose 1; N=390;197) | 14 | 0
  Myalgia (Post-dose 1; N=390;197) | 121 | 52
  Grade 3 Myalgia (Post-dose 1; N=390;197) | 15 | 3
  Asthenia (Post-dose 1; N=390;197) | 77 | 30
  Grade 3 Asthenia (Post dose 1; N=390;197) | 7 | 2
  Fever (Post-dose 2; N=371;184) | 29 | 16
  Grade 3 Fever (Post-dose 2; N=371;184) | 2 | 0
  Headache (Post-dose 2; N=373;185) | 131 | 69
  Grade 3 Headache (Post-dose 2; N=373;185) | 14 | 4
  Malaise (Post-dose 2; N=373;185) | 68 | 36
  Grade 3 Malaise (Post-dose 2; N=373;185) | 6 | 4
  Myalgia (Post dose 2; N=373;185) | 80 | 45
  Grade 3 Myalgia (Post-dose 2; N=373;185) | 8 | 3
  Asthenia (Post-dose 2; N=373;185) | 51 | 24
  Grade 3 Asthenia (Post-dose 2; N=373;185) | 5 | 1
  Fever (Post-dose 3; N=362;180) | 17 | 14
  Grade 3 Fever (Post-dose 3; N=362;180) | 0 | 3
  Headache (Post-dose 3; N=364;180) | 106 | 62
  Grade 3 Headache (Post-dose 3; N=364;180) | 10 | 4
  Malaise (Post-dose 3; N=364;180) | 60 | 41
  Grade 3 Malaise (Post-dose 3; N=364;180) | 2 | 4
  Myalgia (Post-dose 3; N=364;180) | 66 | 51
  Grade 3 Myalgia (Post-dose 3; N=364;180) | 3 | 5
  Asthenia (Post-dose 3; N=364;180) | 42 | 23
  Grade 3 Asthenia (Post-dose 3; N=364;180) | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post vaccination) up to Day 28 after each vaccination.
Arm/Group | Dengue Vaccine Group | Control Group
Serious Adverse Events (participants affected / at risk) | 10/401 | 15/199
Other Adverse Events (participants affected / at risk) | 237/401 | 132/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dengue Vaccine Group (N=401) | Control Group (N=199)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Dengue fever (Infections and infestations) | 3 (3) | 3 (3)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dengue Vaccine Group (N=401) | Control Group (N=199)
Abdominal pain (Gastrointestinal disorders) | 17 (19) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 30 (30) | 9 (10)
Nasopharyngitis (Infections and infestations) | 105 (124) | 51 (61)
Headache (Nervous system disorders) | 35 (40) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 23 (24)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (10)
Injection site Pain (General disorders) | 192/392 (192) | 132/198 (132)
Injection site Erythema (General disorders) | 26/392 (26) | 18/198 (18)
Injection site Swelling (General disorders) | 20/392 (20) | 16/198 (16)
Fever (General disorders) | 84/392 (84) | 36/197 (36)
Headache (Nervous system disorders) | 237/391 (237) | 116/198 (116)
Malaise (General disorders) | 157/390 (157) | 82/198 (82)
Myalgia (Musculoskeletal and connective tissue disorders) | 171/390 (171) | 90/198 (90)
Asthenia (General disorders) | 119/390 (119) | 51/198 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.